CLINICAL TRIAL: NCT00554879
Title: Acupuncture Treatment of Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: Malcolm Grow Medical Clinics and Surgery Center (U.S. Federal Agency)
Responsible Party: Michael J. Mines, Walter Reed Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WU # 07-23024
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Keratoconjunctivitis Sicca; Xeropthalmia
MeSH Terms: conditions — Keratoconjunctivitis Sicca | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Acupuncture
  Interventions: Procedure: Acupuncture
- 2 (Sham Comparator): Sham Acupuncture
  Interventions: Procedure: Sham acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Needles placed bilaterally on the ears at the auriculotherapy points. Additional needles placed in both index fingers. A third set of needles inserted on both index fingers between LI-1 adn LI-2.
  Arms: 1
Procedure: Sham acupuncture — Four needles will be placed on the left and right upper shoulder areas. Small circular adhesive tape will be placed in an ear area, but not on the acupuncture points.
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety and efficacy of acupuncture in the treatment of moderate to severe dry eye by replicating the study design of the previous protocol and to see the study through to its completion.

ELIGIBILITY:
Inclusion Criteria:

* Military healthcare beneficiary
* Male and female patients, at least 18 years of age
* Diagnosis of keratoconjunctivitis sicca or xerophthalmia (dry eyes) in one or both eyes
* Persistent signs and symptoms despite conventional therapy for at least three months

Exclusion Criteria:

* Contact lens wear
* Intraocular surgery or laser in the study eye within 90 days prior to enrolling in the study
* History of any medical condition or circumstance that would preclude scheduled visits or completion of the study
* Known history of adverse reaction to acupuncture
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To answer the question of whether there are objective beneficial effects of an acupuncture treatment versus sham acupuncture on dry eye, as measured by some of the most widely-used clinical indicators in the literature. | 6 months after acupuncture or sham acupuncture treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Mines, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States